CLINICAL TRIAL: NCT06892340
Title: A Non-Invasive, Non-Sedating Device to Mitigate Motion Sickness and Spatial Disorientation
Brief Title: Evaluation of a Device to Reduce Motion Sickness and Spatial Disorientation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Collaborators: Defense Health Agency (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C.2024.076 FWH20240041H; ST 1186 (Other: DHA Restoral / 59th MDW ST)
Record Dates: First submitted 2025-01-17; First posted 2025-03-24 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Motion Sickness
Keywords: Motion Sickness; Simulator Sickness; Trigeminal innervation; Transcutaneous auricular neurostimulation; Sparrow Ascent; Neuromodulation; Simulator adaption syndrome; Transcutaneous vagus nerve stimulation; Auricle; Mild electrical stimulation; Cranial nerves; Occipital nerves; Cymba Concha; Afferent sensory innervation; Vagus Nerve; Auriculotemporal nerve; Trigeminal nerve; Auricular nerve; Cranial nerve V; Cranial nerve VII; Cranial nerve IX; Cranial nerve X; Non-invasive; Non-sedating
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized, double-blinded, sham-controlled investigation of the effects of transcutaneous auricular neurostimulation (tAN) on spatial disorientation and motion sickness. Participants will be recruited from a motion-naïve population and randomized into two groups:
  Group 1 (n = 18): Active tAN initiated 45-minutes before simulated disorientation Group 2 (n = 18): Passive Sham tAN
  Experimentation will take place in 5 stages: (Pre-experimentation)
  1) prior to spatial disorientation challenge, 2) spatial disorientation challenge, 3) between challenges, 4) motion sickness challenge, 5) conclusion
  At the conclusion of pre-experimentation, the subjects will be placed with a tAN earpiece on their left ear. A tAN device will be programmed based on the participant study group and will be connected to the participant's earpiece.
Who Masked: Participant, Investigator
Masking Description: The participants and investigator will be blind to participant treatment group assignment. Only the research coordinator will know the treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sham Transcutaneous Auricular Neurostimulation Device (Group 2) (No Intervention): The Sparrow Ascent Clinical Tool will be used to designate the tAN device as either active or sham. For participants randomized to the sham tAN group (Group 2), the Sparrow Ascent device will be programmed to sham settings. The participant receives a device that is turned on at the time of earpiece placement but does not provide electric stimulation. The subjects will remain blinded to their group assignment. At each interaction with the subject, the research coordinator will inform the subject that the device may be activated, and they may or may not feel stimulation at the time of activation.
  Subjects will then undergo spatial disorientation and motion sickness challenges. Vital signs will be obtained at specific time markers, and questionnaires and assessments completed.
- Active Transcutaneous Auricular Neurostimulator Device (Group 1) (Active Comparator): The Sparrow Ascent Clinical Tool will be used to designate the tAN device as either active or sham. For participants randomized to the active tAN group (Group 1), the Sparrow Ascent device will be programmed to the preset stimulation parameters. If the participant states that the stimulation intensity is discomforting, the research coordinator will gradually decrease/increase until a comfortable stimulation intensity is achieved. After the device is programmed, participants' stimulation amplitude (in mA) will be documented.
  The subjects will remain blinded to their group assignment. At each interaction with the subject, the research coordinator will inform the subject that the device may be activated, and they may or may not feel stimulation at the time of activation.
  Subjects will then undergo spatial disorientation and motion sickness challenges. Vital signs will be obtained at specific time markers, and questionnaires and assessments completed.
  Interventions: Device: Transcutaneous Auricular Neurostimulation device

INTERVENTIONS:
Device: Transcutaneous Auricular Neurostimulation device — The Sparrow Ascent device will be programmed to the preset stimulation parameters. Two individual stimulation frequencies will be set: 15 Hz at cymba concha (Region 1/Channel 1; vagal innervation) and 100 Hz adjacently anterior to the tragus (Region 2/Channel 2; trigeminal innervation). The pulse duration will be set to 250 #s for all participants. The stimulation intensities (mA) will be set to 1.0 and 1.4 (for Region 1 and 2, respectively) based on the median values observed in the previous data set. If the participant states that the stimulation intensity is discomforting, the research coordinator will gradually decrease/increase until a comfortable stimulation intensity is achieved
  Arms: Active Transcutaneous Auricular Neurostimulator Device (Group 1)

SUMMARY:
The purpose of this research study is to learn how a wearable nerve stimulation device, the Spark Biomedical's Sparrow Ascent System™, impacts the development of spatial disorientation and/or motion sickness in a healthy population.

Spatial disorientation is when there is a "mismatch" between where a person is, and where the sense organs in their body tell them where they are. These sense organs include the inner ear (the vestibular system), the eyes (the visual system), the sense of where one's legs, back, and neck are (proprioceptive system), and one's higher thinking (cognitive centers). If spatial disorientation is severe or occurs in motion-naïve individuals, spatial disorientation can lead to motion sickness.

The Sparrow Ascent System™ is a wearable, battery-operated transcutaneous auricular (ear) neurostimulation (tAN) device. This means that it uses electrical pulses to stimulate branches of nerves on and/or around the ear, specifically the "vagus" and "trigeminal" nerves. These nerves are also responsible for your sensation of nausea and your heart rate (vagus nerve), as well as headaches (trigeminal nerve). The Sparrow System utilizes a flexible earpiece with embedded hydrogel electrodes that stick to the skin, the earpiece is disposable after use. This device is already Food and Drug Administration (FDA) approved for use in humans and is safely used for control of symptoms in a variety of other medical conditions, such as opioid withdrawal and acute stress reaction. In this study, we will determine if the Sparrow Ascent System™ impacts the development of spatial disorientation or motion sickness.

DETAILED DESCRIPTION:
The purpose of this research study is to learn how a wearable nerve stimulation device, the Spark Biomedical's Sparrow Ascent System™, impacts the development of spatial disorientation and/or motion sickness in a healthy population. Study participants will be given monitoring equipment to wear during the study, which will record the participant's vital signs throughout the experiment.

Participants will be randomly assigned to one of two groups. Randomization is a process like flipping a coin and meaning there is a chance of being assigned to either of the groups. The two groups include one group where the Sparrow Ascent System™ is turned on. The second group will be given a "sham" Sparrow Ascent System™. A sham device is an inactive Spark Sparrow Therapy System™ that looks like the normal device, but that does not provide any therapy.

Participants will be given different stimuli that may cause spatial disorientation and motion sickness. This will include an electronic flight simulator and a rotating chair. In the flight simulator, participants will be given different tasks to complete that often cause some minor spatial disorientation. In the rotating chair, investigators will spin participants around at a steady rate for 10 minutes and ask the participants to change the participants head position in ways that often cause motion sickness. Before, during, and after these stimuli participants will be asked to complete a series of tests to determine if the participants are becoming susceptible to either spatial disorientation or motion sickness. These tests will include asking how the participants are feeling throughout the stimuli, written questionnaires about how the participants feel. Before and after stimuli, participants will also be asked to perform simple tasks to test the participants orientation and performance including hand-eye-coordination, object tracking, and reaction time.

ELIGIBILITY:
* Inclusion Criteria:

  1. Healthy males and non-pregnant females between the ages of 18-50 who do not experience symptoms of motion sickness.
  2. Participants who are English speaking.
  3. Participants who are able to read and understand study procedures in order to provide informed consent.
* Exclusion Criteria:

  1. Females who are pregnant
  2. Cardiac pathology (congestive heart failure, history of myocardial infarction, cardiac stent placement, pacemaker placement, heart surgery)
  3. Hypertension requiring daily medication
  4. Active vestibular disease to include Meniere's disease, migraine associated vertigo, benign paroxysmal positional vertigo, labyrinthitis
  5. Neck pain or spinal pathology
  6. Medications impacting cardiac, vestibular, or neurologic function
  7. Recently ill or hospitalized within 30 days
  8. Pilots and individuals formally desensitized to motion sickness
  9. Use of vestibular suppressing medications or drugs within 24 hours of the study (antihistamines, histamine-1 receptor agonists, benzodiazepines, anticholinergics, dopamine receptor agonists, alcohol, marijuana, tobacco, opiates)
  10. Participant has a history of epileptic seizures
  11. Participant has a history of neurological diseases or traumatic brain injury
  12. Abnormal vital signs obtained during pre-experimentation phase:
* Heart Rate >100 or <50
* Systolic blood pressure >150 or <90
* Respiratory rate >24 or <8 13. Participant has presence of devices, e.g., pacemakers, cochlear prosthesis, neurostimulators 14. Participant has abnormal ear anatomy or ear infection present 15. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Graybiel Scale | Baseline, and at 5- and 10-minutes post motion sickness and at 5- and 10-minutes post spatial disorientation challenges.
  The Graybiel scale is a commonly used scale for identifying and rating motion sickness symptoms. It was designed to survey multiple dimensions of motion sickness characterized by the degree of 6 representative cardinal symptoms: Nausea and vomiting, skin color, cold sweating, increased salivation, drowsiness, pain and central nervous system symptoms. Each cardinal symptom category is rated by the participant and a corresponding score is calculated. Lesser symptoms are scored with lower point values, 1, 2 or 4 points depending on the severity of that particular symptom with higher scores indicating increased severity. More severe symptoms are scored 8 or 16 points. Values greater than or equal to 16 total points is categorized as frank sickness, 8 to 15 points is severe malaise, 5 to 7 points is moderate malaise A, 3 to 4 points is moderate malaise B, and 1 to 2 points is categorized as slight malaise.

SECONDARY OUTCOMES:
Vitals: Blood pressure | Baseline and immediately post spatial disorientation challenge and immediately post motion sickness challenge. At 90 minutes post motion sickness challenge.
  The force of blood pushing against the walls of arteries. Two pressures are measured in mm Hg and are captured via a blood pressure cuff. The systolic pressure in the arteries when the heart contracts and the diastolic pressure in the arteries when the heart relaxes. This is shown numerically with the systolic pressure over the diastolic pressure.
Misery Scale (MISC) | Baseline, and at 3 times during the spatial disorientation challenge, at 5- and 10-minutes post spatial disorientation challenge as well as 1-minute intervals during the motion sickness challenge and 5- and 10-minutes post motion sickness challenge.
  Misery Scale (MISC); an 11-point rating scale used to measure the severity of motion sickness symptoms, ranging from no symptoms at all (0) to severe nausea and vomiting (10), with intermediate levels representing increasing discomfort. It measures how "miserable" one feels due to motion sickness. It provides a detailed progression of symptoms to better understand the severity of motion sickness.
Motion Sickness Assessment Questionnaire (MSAQ) | Baseline, and 5- and 10-minutes post spatial disorientation challenge and 5- and 10-minutes post motion sickness challenge.
  Motion Sickness Assessment Questionnaire (MSAQ). An instrument that helps assess the experience of motion sickness on a multi-dimensional level. The MSAQ measures four dimensions of motion sickness, gastrointestinal, central, peripheral, and sopite-related (drowsiness, yawning, disengagement). Motion sickness can be a complex set of interacting psychophysiological symptoms that are hard to define. Moreover, one person may experience one symptom to a greater degree than another person, yet both would be experiencing "motion sickness". Additionally, an individual may experience a different feeling of motion sickness depending on the context of what is causing the motion sickness, (boat vs. vehicle vs. visual stimulus) with each potentially eliciting different symptoms. Participants are asked to assess their motion sickness experience by rating 16 statements (ex. I felt sick to my stomach, I felt faint like) from 1-9 with increasing numbers indicating increased severity.
Simulator sickness questionnaire (SSQ) | Baseline and at 5- and 10-minutes post spatial disorientation challenge and 5- and 10-minutes post motion sickness challenge.
  The Simulator Sickness Questionnaire (SSQ), a tool that helps assess the effects of the environment on an individual's health. A set of sixteen symptoms qualified under nausea, oculomotor discomfort, and disorientation categories are rated from one to four from (1 none, 2 slight, 3 moderate, 4 severe). These symptoms include general discomfort, fatigue, headache, eye strain, difficulty focusing, increased salivation, sweating, nausea, difficulty concentrating, fullness of head, blurred vision, dizzy (eyes open), dizzy (eyes closed), vertigo, stomach awareness and burping. Via calculations the answer to each symptom specific severity question results in three representative sub scores, Nausea related, Oculomotor related, and Disorientation related. These are then combined to get an overall simulator sickness severity score. The SSQ was developed in response to motion sickness questionnaires being deficient or irrelevant in measuring simulator sickness.
Motion sickness susceptibility questionnaire | Baseline
  The Motion sickness Susceptibility Questionnaire predicts individual differences in motion sickness based on stimuli. This questionnaire considers motion type (cars, fair rides, trains, planes etc.), sickness severity ratings, childhood versus adult experiences to find out how susceptible an individual may be to motion sickness and what sorts of motion are the most effective in causing sickness. The participant is asked to rate each motion type as never felt sick, rarely felt sick, sometimes felt sick, frequently felt sick or not applicable if they never traveled via that particular motion type. They are asked the same questions for "As a child" and "Over the last 10 years".
Functional Ability Assessment | Baseline and 15 minutes post spatial disorientation challenge and 15 minutes post motion sickness challenge.
  The Senaptec Sensory Station is a state-of-art sensory evaluation & training station which assesses 10 visual and sensorimotor skills including visual clarity, contrast sensitivity, depth perception, near-far quickness, perception span, multiple object tracking, reaction time, target capture, eye-hand coordination and go / no go. This assessment will give the study team a baseline reference for the subject's functional ability which will then be compared/contrasted to the same assessment given post each spatial disorientation and motion sickness challenge.
Vitals: Heart rate | Continuously throughout the study day, starting at baseline and stopping 90 minutes post motion sickness challenge.
  The number of times a person's heart beats in one minute. Source: Polar H10 Heart Rate Sensor.
Vitals: Heart Rate Variability | Continuously throughout the study day, starting at baseline and stopping 90 minutes post motion sickness challenge.
  Heart rate variability is the variation in time between heart beats. It is a measure of how well your body can handle stress and recover from physical activity. Source: Polar H10 Heart Rate Sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac D Erbele, MD, ENT, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Randolph AFB Physiology lab, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication to 6 years after publication.
Access Criteria: Researchers may contact the principal investigator for access. Available data will include subject demographics, study group, and instruments values.

REFERENCES:
- [Background] Heinle, Todd E. and William R. Ercoline. "Spatial Disorientation: Causes, Consequences and Countermeasures for the USAF." (2003).
- [Background] Mark S. George, Ziad Nahas, Daryl E. Bohning, Qiwen Mu, F. Andrew Kozel, Jeffrey Borckhardt, Stewart Denslow, Mechanisms of action of vagus nerve stimulation (VNS), Clinical Neuroscience Research, Volume 4, Issues 1-2, 2004, Pages 71-79, ISSN 1566-2772, https://doi.org/10.1016/j.cnr.2004.06.006.
- [Background] Ebenholtz SM, Cohen MM, Linder BJ. The possible role of nystagmus in motion sickness: a hypothesis. Aviat Space Environ Med. 1994 Nov;65(11):1032-5. PMID 7840743
- [Background] Rogers D, Van Syoc D. Clinical Practice Guideline for Motion Sickness. November 2011. http://www.asams. org/guidelines/Completed/NEW%20Motion%20Sickness.htm. Accessed January 11, 2022.
- [Background] Kramer MR, Wasserman EB, Teel EF, et al Effect of protective helmets on vision and sensory performance. British Journal of Sports Medicine 2017;51:A65.
- [Background] Caserman, P., Garcia-Agundez, A., Gámez Zerban, A. et al. Cybersickness in current-generation virtual reality head-mounted displays: systematic review and outlook. Virtual Reality 25, 1153-1170 (2021). https://doi.org/10.1007/s10055-021-00513-6
- [Background] Chan G, Moochhala SM, Zhao B, Wl Y, Wong J. A comparison of motion sickness prevalence between seafarers and non-seafarers onboard naval platforms. Int Marit Health. 2006;57(1-4):56-65. PMID 17312694
- [Background] Antunano MJ, Hernandez JM. Incidence of airsickness among military parachutists. Aviat Space Environ Med. 1989 Aug;60(8):792-7. PMID 2775137
- [Background] Jenkins DD, Khodaparast N, O'Leary GH, Washburn SN, Covalin A, Badran BW. Transcutaneous Auricular Neurostimulation (tAN): A Novel Adjuvant Treatment in Neonatal Opioid Withdrawal Syndrome. Front Hum Neurosci. 2021 Mar 8;15:648556. doi: 10.3389/fnhum.2021.648556. eCollection 2021. PMID 33762918
- [Background] Tirado CF, Washburn SN, Covalin A, Hedenberg C, Vanderpool H, Benner C, Powell DP, McWade MA, Khodaparast N. Delivering transcutaneous auricular neurostimulation (tAN) to improve symptoms associated with opioid withdrawal: results from a prospective clinical trial. Bioelectron Med. 2022 Aug 18;8(1):12. doi: 10.1186/s42234-022-00095-x. PMID 35978394
- [Background] Cowings PS, Toscano WB, DeRoshia C, Tauso R. Effects of Command and Control Vehicle (C2V) operational environment on soldier health and performance. Hum Perf Extrem Environ. 2001 Jun;5(2):66-91. PMID 14649629
- [Background] Molefi E, McLoughlin I, Palaniappan R. On the potential of transauricular electrical stimulation to reduce visually induced motion sickness. Sci Rep. 2023 Feb 25;13(1):3272. doi: 10.1038/s41598-023-29765-9. PMID 36841838
- [Background] Bauer S, Baier H, Baumgartner C, Bohlmann K, Fauser S, Graf W, Hillenbrand B, Hirsch M, Last C, Lerche H, Mayer T, Schulze-Bonhage A, Steinhoff BJ, Weber Y, Hartlep A, Rosenow F, Hamer HM. Transcutaneous Vagus Nerve Stimulation (tVNS) for Treatment of Drug-Resistant Epilepsy: A Randomized, Double-Blind Clinical Trial (cMPsE02). Brain Stimul. 2016 May-Jun;9(3):356-363. doi: 10.1016/j.brs.2015.11.003. Epub 2016 Jan 20. PMID 27033012
- [Background] McIntire LK, McKinley RA, Goodyear C, McIntire JP, Brown RD. Cervical transcutaneous vagal nerve stimulation (ctVNS) improves human cognitive performance under sleep deprivation stress. Commun Biol. 2021 Jun 10;4(1):634. doi: 10.1038/s42003-021-02145-7. PMID 34112935
- [Background] Yakunina N, Kim SS, Nam EC. Optimization of Transcutaneous Vagus Nerve Stimulation Using Functional MRI. Neuromodulation. 2017 Apr;20(3):290-300. doi: 10.1111/ner.12541. Epub 2016 Nov 29. PMID 27898202
- [Background] Frangos E, Ellrich J, Komisaruk BR. Non-invasive Access to the Vagus Nerve Central Projections via Electrical Stimulation of the External Ear: fMRI Evidence in Humans. Brain Stimul. 2015 May-Jun;8(3):624-36. doi: 10.1016/j.brs.2014.11.018. Epub 2014 Dec 6. PMID 25573069
- [Background] Badran BW, Dowdle LT, Mithoefer OJ, LaBate NT, Coatsworth J, Brown JC, DeVries WH, Austelle CW, McTeague LM, George MS. Neurophysiologic effects of transcutaneous auricular vagus nerve stimulation (taVNS) via electrical stimulation of the tragus: A concurrent taVNS/fMRI study and review. Brain Stimul. 2018 May-Jun;11(3):492-500. doi: 10.1016/j.brs.2017.12.009. Epub 2017 Dec 29. PMID 29361441
- [Background] Babic T, Browning KN. The role of vagal neurocircuits in the regulation of nausea and vomiting. Eur J Pharmacol. 2014 Jan 5;722:38-47. doi: 10.1016/j.ejphar.2013.08.047. Epub 2013 Oct 31. PMID 24184670
- [Background] Suzuki T, Sugiyama Y, Yates BJ. Integrative responses of neurons in parabrachial nuclei to a nauseogenic gastrointestinal stimulus and vestibular stimulation in vertical planes. Am J Physiol Regul Integr Comp Physiol. 2012 Apr 15;302(8):R965-75. doi: 10.1152/ajpregu.00680.2011. Epub 2012 Jan 25. PMID 22277934
- [Background] Balaban CD. Projections from the parabrachial nucleus to the vestibular nuclei: potential substrates for autonomic and limbic influences on vestibular responses. Brain Res. 2004 Jan 16;996(1):126-37. doi: 10.1016/j.brainres.2003.10.026. PMID 14670639
- [Background] Zhao Q, Ning BF, Zhou JY, Wang J, Yao YJ, Peng ZY, Yuan ZL, Chen JDZ, Xie WF. Transcutaneous Electrical Acustimulation Ameliorates Motion Sickness Induced by Rotary Chair in Healthy Subjects: A Prospective Randomized Crossover Study. Neuromodulation. 2022 Dec;25(8):1421-1430. doi: 10.1016/j.neurom.2021.09.004. Epub 2021 Dec 18. PMID 35088725
- [Background] Eren OE, Filippopulos F, Sonmez K, Mohwald K, Straube A, Schoberl F. Non-invasive vagus nerve stimulation significantly improves quality of life in patients with persistent postural-perceptual dizziness. J Neurol. 2018 Oct;265(Suppl 1):63-69. doi: 10.1007/s00415-018-8894-8. Epub 2018 May 21. PMID 29785522
- [Background] Muth ER. Motion and space sickness: intestinal and autonomic correlates. Auton Neurosci. 2006 Oct 30;129(1-2):58-66. doi: 10.1016/j.autneu.2006.07.020. Epub 2006 Sep 6. PMID 16950658